CLINICAL TRIAL: NCT02944266
Title: Focussed Echocardiography to Detect Preoperative Hypovolemia and Left Ventricular Dysfunction as a Predictor of Post-Induction Hypotension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, J S Rahul, Junior resident , Department of Anaesthesia and Intensive care, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: NK/2172/MD/11249-50
Record Dates: First submitted 2016-10-13; First posted 2016-10-25 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Hypotension
Keywords: post general anaesthesia induced
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hypovolemia group: Those patients who are said to be positive for one or more of the following TTE criteria are grouped under this , them being i.IVC diameter of less than 1 cm , ii.Caval index of > 50%, iii.Left ventricular end diastolic area of < 10 cm2 iv. VTI variation with respiration of < 12.5%, are grouped under the hypovolaemia group .
  Interventions: Other: Pre operative Focus assessed Transthoracic echocardiographic assessment.
- Normovolaemia group: Those patients without the above said TTE findings are hypothesised to be normovolaemic and grouped in here.
  Interventions: Other: Pre operative Focus assessed Transthoracic echocardiographic assessment.

INTERVENTIONS:
Other: Pre operative Focus assessed Transthoracic echocardiographic assessment.

SUMMARY:
This is an observational study to evaluate the role of a Bed side Focus assessed Transthoracic Echocardiography (FATE) in identifying the patients at a potential risk of developing hypotension secondary to general anesthesia induction using the FATE parameters like velocity time integral ( VTI ), Inferior venacava diameter , Caval index and Left ventricular end end diastolic area.

DETAILED DESCRIPTION:
Various haemodynamic parameters like central venous pressure , pulmonary capillary wedge pressure , systolic pulse pressure variations , stroke volume variation , pleth variability index etc are being used as markers of volume status and which in turn have been used as indicators of post general anesthesia induction hypotension in the past . In the current study the investigators aim to validate the role of a bed side 2-D transthoracic echocardiography (TTE) as a guide to identify the volume status of the patient before induction and clinically observe for the haemodynamic changes in the form of mean arterial pressure variations in the immediate post induction period.

The investigators aim to perform preoperative bed side Transthoracic echocardiography in 150 American society of Anesthesiologists grade-I/II patients posted for routine General anaesthesia procedures and assess their volume status . Then the investigators would collect 10 mean arterial pressure recordings at one minute interval in the immediate postinduction period and assess the accuracy of TTE in identifying potential patients at risk of developing post induction hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Any ASA - I/II patient posted for a routine general anaesthesia procedure and who do not fit with the exclusion criteria.

Exclusion Criteria:

* a) Extremes of age <18 years and >60 years

  b) BMI<18 and >40

  c) Patients with pre-existing hemodynamic instability, ventricular dysfunction and

Sepsis.

d) Patients on beta blocking agents.

e) Preinduction mean arterial pressure of <70 mm hg.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Any ASA - I/II patient posted for a routine general anaesthesia procedure who is between the age groups 18-60 years, with a BMI between 18-40 , without preexisting haemodynamic instability , sepsis or a documented ventricular dysfunction.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Focussed Echocardiography to Detect Preoperative Hypovolemia and Left Ventricular Dysfunction as a Predictor of Post-Induction Hypotension | January 2016- November 2016
  Role of Transthoracic echocardiography in assessing preoperative volume status using various parameters like Velocity time integral , Inferior vena cava diameter , Caval index , Left Ventricular end diastolic area etc ., in accurately predicting the incidence of hypotension at the time of induction in patients who are being administered general anaesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- J S Rahul, Chandigarh, Chandigarh, India

REFERENCES:
- [Background] Reich DL, Hossain S, Krol M, Baez B, Patel P, Bernstein A, Bodian CA. Predictors of hypotension after induction of general anesthesia. Anesth Analg. 2005 Sep;101(3):622-628. doi: 10.1213/01.ANE.0000175214.38450.91. PMID 16115962
- [Background] Lienhart A, Auroy Y, Pequignot F, Benhamou D, Warszawski J, Bovet M, Jougla E. Survey of anesthesia-related mortality in France. Anesthesiology. 2006 Dec;105(6):1087-97. doi: 10.1097/00000542-200612000-00008. PMID 17122571
- [Background] Devereaux PJ, Goldman L, Cook DJ, Gilbert K, Leslie K, Guyatt GH. Perioperative cardiac events in patients undergoing noncardiac surgery: a review of the magnitude of the problem, the pathophysiology of the events and methods to estimate and communicate risk. CMAJ. 2005 Sep 13;173(6):627-34. doi: 10.1503/cmaj.050011. PMID 16157727
- [Background] Bijker JB, van Klei WA, Vergouwe Y, Eleveld DJ, van Wolfswinkel L, Moons KG, Kalkman CJ. Intraoperative hypotension and 1-year mortality after noncardiac surgery. Anesthesiology. 2009 Dec;111(6):1217-26. doi: 10.1097/ALN.0b013e3181c14930. PMID 19934864
- [Background] Michard F, Teboul JL. Predicting fluid responsiveness in ICU patients: a critical analysis of the evidence. Chest. 2002 Jun;121(6):2000-8. doi: 10.1378/chest.121.6.2000. PMID 12065368
- [Background] Michard F. Changes in arterial pressure during mechanical ventilation. Anesthesiology. 2005 Aug;103(2):419-28; quiz 449-5. doi: 10.1097/00000542-200508000-00026. PMID 16052125
- [Background] Feissel M, Michard F, Faller JP, Teboul JL. The respiratory variation in inferior vena cava diameter as a guide to fluid therapy. Intensive Care Med. 2004 Sep;30(9):1834-7. doi: 10.1007/s00134-004-2233-5. Epub 2004 Mar 25. PMID 15045170
- [Background] Reuter DA, Felbinger TW, Schmidt C, Kilger E, Goedje O, Lamm P, Goetz AE. Stroke volume variations for assessment of cardiac responsiveness to volume loading in mechanically ventilated patients after cardiac surgery. Intensive Care Med. 2002 Apr;28(4):392-8. doi: 10.1007/s00134-002-1211-z. Epub 2002 Mar 20. PMID 11967591
- [Background] Feissel M, Michard F, Mangin I, Ruyer O, Faller JP, Teboul JL. Respiratory changes in aortic blood velocity as an indicator of fluid responsiveness in ventilated patients with septic shock. Chest. 2001 Mar;119(3):867-73. doi: 10.1378/chest.119.3.867. PMID 11243970
- [Background] Filipovic M, Seeberger MD, Schneider MC, Schmid M, Pargger H, Hunziker P, Skarvan K. Transthoracic echocardiography for perioperative haemodynamic monitoring. Br J Anaesth. 2000 Jun;84(6):800-3. doi: 10.1093/oxfordjournals.bja.a013596. PMID 10895760
- [Background] Jensen MB, Sloth E, Larsen KM, Schmidt MB. Transthoracic echocardiography for cardiopulmonary monitoring in intensive care. Eur J Anaesthesiol. 2004 Sep;21(9):700-7. doi: 10.1017/s0265021504009068. PMID 15595582
- [Background] Cowie B. Focused cardiovascular ultrasound performed by anesthesiologists in the perioperative period: feasible and alters patient management. J Cardiothorac Vasc Anesth. 2009 Aug;23(4):450-6. doi: 10.1053/j.jvca.2009.01.018. Epub 2009 Mar 19. PMID 19303330
- [Background] American Society of Anesthesiologists and Society of Cardiovascular Anesthesiologists Task Force on Transesophageal Echocardiography. Practice guidelines for perioperative transesophageal echocardiography. An updated report by the American Society of Anesthesiologists and the Society of Cardiovascular Anesthesiologists Task Force on Transesophageal Echocardiography. Anesthesiology. 2010 May;112(5):1084-96. doi: 10.1097/ALN.0b013e3181c51e90. No abstract available. PMID 20418689
- [Background] Colreavy FB, Donovan K, Lee KY, Weekes J. Transesophageal echocardiography in critically ill patients. Crit Care Med. 2002 May;30(5):989-96. doi: 10.1097/00003246-200205000-00007. PMID 12006793
- [Background] Brienza N, Giglio MT, Marucci M, Fiore T. Does perioperative hemodynamic optimization protect renal function in surgical patients? A meta-analytic study. Crit Care Med. 2009 Jun;37(6):2079-90. doi: 10.1097/CCM.0b013e3181a00a43. PMID 19384211
- [Background] Alecu C, Cuignet-Royer E, Mertes PM, Salvi P, Vespignani H, Lambert M, Bouaziz H, Benetos A. Pre-existing arterial stiffness can predict hypotension during induction of anaesthesia in the elderly. Br J Anaesth. 2010 Nov;105(5):583-8. doi: 10.1093/bja/aeq231. Epub 2010 Aug 26. PMID 20798172
- [Background] Tsuchiya M, Yamada T, Asada A. Pleth variability index predicts hypotension during anesthesia induction. Acta Anaesthesiol Scand. 2010 May;54(5):596-602. doi: 10.1111/j.1399-6576.2010.02225.x. Epub 2010 Mar 10. PMID 20236098
- [Background] Shillcutt SK, Markin NW, Montzingo CR, Brakke TR. Use of rapid "rescue" perioperative echocardiography to improve outcomes after hemodynamic instability in noncardiac surgical patients. J Cardiothorac Vasc Anesth. 2012 Jun;26(3):362-70. doi: 10.1053/j.jvca.2011.09.029. Epub 2012 Jan 4. PMID 22226417
- [Background] Gauss A, Heinrich H, Wilder-Smith OH. Echocardiographic assessment of the haemodynamic effects of propofol: a comparison with etomidate and thiopentone. Anaesthesia. 1991 Feb;46(2):99-105. doi: 10.1111/j.1365-2044.1991.tb09349.x. PMID 1872460
- [Background] Mulier JP, Wouters PF, Van Aken H, Vermaut G, Vandermeersch E. Cardiodynamic effects of propofol in comparison with thiopental: assessment with a transesophageal echocardiographic approach. Anesth Analg. 1991 Jan;72(1):28-35. doi: 10.1213/00000539-199101000-00006. PMID 1984373
- [Background] Mackenzie DC, Noble VE. Assessing volume status and fluid responsiveness in the emergency department. Clin Exp Emerg Med. 2014 Dec 31;1(2):67-77. doi: 10.15441/ceem.14.040. eCollection 2014 Dec. PMID 27752556